CLINICAL TRIAL: NCT07009600
Title: Impact of Targeted Therapy and Immune Checkpoint Inhibitors on Prognosis and Surgical Outcomes in Conversion Surgery for Stage IV Gastric Cancer
Brief Title: Conversion Surgery After Target Therapy or Immunotherapy in Stage IV Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung Eun Oh, Clinical assistant professor, Samsung Medical Center
Other Study IDs: SMC 2025-03-046-001
Record Dates: First submitted 2025-05-23; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors; Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: immune check point inhibitors (PD-1 inhibitors), target therapy (trastuzumab)

SUMMARY:
In this retrospective study, investigators conducted a comprehensive investigation of the factors influencing postoperative prognosis in patients with stage IV gastric cancer undergoing conversion surgery. Specifically, investigators examined the impact of targeted therapy or immune check point inhibitors (ICIs) in combination with preoperative chemotherapy on (1) prognostic differences based on initial progression (invading adjacent organs) and metastatic site (peritoneum, distant lymph node [LN]) at the time of stage IV gastric cancer diagnosis and (2) conversion surgery outcomes and pathological complete response (pCR).

ELIGIBILITY:
Inclusion Criteria:

* Stage IV gastric cancer patients who underwent conversion surgery

Exclusion Criteria:

* Patients who did not undergo gastrectomy
* Patients who underwent emergent surgery due to cancer perforation
* Patients with missing medical records or information

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically diagnosed and histologically confirmed stage IV gastric cancer between January 2010 and August 2024 and received systemic palliative-intent chemotherapy as initial treatment and underwent conversion surgery at Samsung Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
overall survival and disease free survival | from date of surgery until the date of first documented cancer recurrence or date of death from cancer progression, whichever came first, assessed up to 160 months